CLINICAL TRIAL: NCT04917198
Title: Median Sternotomy in Penetrating Cardiac Trauma Does it Make a Difference?
Brief Title: Median Sternotomy in Penetrating Cardiac Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Ibrahim Gadallah, Median sternotomy in penetrating cardiac trauma , does it make a difference?, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Median sternotomy
Record Dates: First submitted 2021-05-20; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Trauma Chest
MeSH Terms: conditions — Thoracic Injuries | interventions — Sternotomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- median sternotomy (Experimental): median sternotomy in penetrating cardiac trauma and hemodynamically unstable patients, does it affect morbidity and mortality.
  Interventions: Procedure: median sternotomy

INTERVENTIONS:
Procedure: median sternotomy — median sternotomy

SUMMARY:
The investigators aim to assess role of median sternotomy in penetrating cardiac trauma regarding morbidity and mortality of the patients.

DETAILED DESCRIPTION:
Cardiac trauma is a leading cause of death in the USA and occurs mostly due to motor vehicle accidents. Cardiac trauma may be blunt or as a penetrating chest injuries, and both can lead to aortic injuries. The Right Ventricle followed by the Left Ventricle was the most common site of injury.

Timely diagnosis and early management are the key to improve mortality. Mortality related to cardiac trauma remains high despite improvement in diagnosis and management.

Assessment of suspected cardiac injuries in a trauma setting is a challenging and time-critical matter, with clinical and imaging findings having complementary roles in the formation of an accurate diagnosis. Cardiac computed tomography and cardiac ultrasound are the two most important diagnostic modalities.

Pericardial tamponade and haemothorax were common intra-operative findings. Patients having penetrating cardiac injury presenting with detectable signs of life on arrival to the hospital can be rescued by early surgical intervention.

Penetrating cardiac injuries are high-risk, high-mortality injuries considering the outcomes. Therefore, it is important to choose the appropriate incision. In general clinical settings, thoracotomy and median sternotomy are choices of incisions to explore the injury.

It is really important to transfer these patients to the nearest facility in time, make sure they get immediate diagnosis and proper resuscitation until they are ready to be taken into the operating room for exploration.

ELIGIBILITY:
Inclusion Criteria:

* A. Inclusion criteria:

Penetrating traumatic cardiac patients. B.age:patients aged from15 to 60 years old.

Exclusion Criteria:

* Patient who arrest immediately when arrived trauma unit.
* patients with polytrauma
* patients with chronic medical disease as asthma or ischemic herat disease

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-21 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Time needed to explore heart | baseline
  To reveal time needed to explore heart in both interventions.

SECONDARY OUTCOMES:
Pain by pain score | baseline
  Post operative pain complained by patient.

REFERENCES:
- [Background] Gosavi S, Tyroch AH, Mukherjee D. Cardiac Trauma. Angiology. 2016 Nov;67(10):896-901. doi: 10.1177/0003319715627954. Epub 2016 Jul 11. PMID 26802100
- [Background] Leite L, Goncalves L, Nuno Vieira D. Cardiac injuries caused by trauma: Review and case reports. J Forensic Leg Med. 2017 Nov;52:30-34. doi: 10.1016/j.jflm.2017.08.013. Epub 2017 Aug 24. PMID 28850860
- [Background] Rahim Khan HA, Gilani JA, Pervez MB, Hashmi S, Hasan S. Penetrating cardiac trauma: A retrospective case series from Karachi. J Pak Med Assoc. 2018 Aug;68(8):1285-1287. PMID 30108408